CLINICAL TRIAL: NCT01502865
Title: Clinician Access to Soldier Suicide Information (CASSI)
Acronym: CASSI
Status: Withdrawn | Type: Observational
Why Stopped: Should not have been listed on ClinicalTrials
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter M. Gutierrez, Clincial/Research Psychologist, VA Eastern Colorado Health Care System
Other Study IDs: COMIRB 10-1168
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this project is to conduct a feasibility study using data proved by Department of Defense National Center for Telehealth and Technology (T2) toward the ultimate goal of establishing a mechanism by which VA clinicians could access data on Veterans regarding suicidal thoughts and/or behaviors that occurred when they were on active duty, as documented in the Department of Defense Suicide Event Report (DoDSER).

DETAILED DESCRIPTION:
As a first step toward the overall goal of this project, the investigators will use data from T2 to conduct the first stage of a feasibility study. Specifically, the investigators will attempt to match Social Security numbers (SSNs) of Soldiers who have had suicidal thoughts and/or behaviors in the DoDSER against SSNs of Veterans seeking mental health services at any VA in the United States. Once this first step has been accomplished, the investigators also aim to describe the group of Veterans with DoDSERs who are accessing VA services (i.e., demographic information, military service variables, and health care utilization variables) in an attempt to better understand this group. It is anticipated that if this study is successful, a next step would be to explore the possibility of DoDSER data sharing with VA partners toward attainment of the following long-term goals: 1. Sharing information on history of active duty suicidal thoughts and/or behaviors among discharged individuals seeking mental health services in VA systems; 2. Facilitating identification of these Veterans; 3. Reducing VA clinician burden though effective access to existing data that may help in assessment and treatment planning; 4. Lowering health care costs through effective early management; 5. Improving quality of care for Veterans seeking services through VA outpatient mental health clinics.

ELIGIBILITY:
Inclusion Criteria:

* Identified with a history of suicidal thoughts and/or behaviors, as recorded in the Army DoDSER

Exclusion Criteria:

* Death by suicide contained in the Army DoDSER (i.e., this information will not be sent to us by T2)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: As of December 2009, there were 6,901 non-fatal Department of Defense Suicide Event Reports(DoDSERs) available for comparison to the VA system. The investigators propose to analyze up to 8,500 that may be available for analysis by the time the protocol is approved.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Gutierrez, PhD, Principal Investigator — VA VISN 19 MIRECC
Locations (1):
- VISN 19 Mental Illness Research Education and Clinical Center, Denver, Colorado, United States

REFERENCES:
- See also: Related Info — http://www.mirecc.va.gov/visn19/